CLINICAL TRIAL: NCT07197749
Title: Administration of Vitamin C (Ascorbic Acid) With Steroids for First Line Therapy of Gastrointestinal GVHD
Brief Title: Vitamin C With Steroids for Gastrointestinal GVHD
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, LaQuisa Hill, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-58040 Vit C for GVHD
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Graft-versus-host-disease (GVHD); Gastrointestinal
Keywords: Graft-Versus-Host-Disease; GVHD; Vitamin C; Gastrointestinal
MeSH Terms: conditions — Graft vs Host Disease | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Patients will be treated with intravenous (IV) or oral (PO) vitamin C depending on the severity of symptoms, ability to tolerate PO intake, and location of treatment (inpatient versus outpatient setting).
  Interventions: Drug: Vitamin C (Ascorbic Acid)

INTERVENTIONS:
Drug: Vitamin C (Ascorbic Acid) — All patients enrolled on this trial will receive steroids at a minimum dose of prednisone 2 mg/kg/day PO (or methylprednisolone 1.6 mg/kg/day IV) divided into 1-2 daily doses as therapy for acute GVHD. For patients that weigh over 100 kg, maximal starting dose of prednisone will be 200 mg (or methylprednisolone-equivalent).
  Patients will be treated with intravenous (IV) or oral (PO) vitamin C depending on the severity of symptoms, ability to tolerate PO intake, and location of treatment (inpatient versus outpatient setting): IV dosing:
  50 mg/kg/day divided TID (max 4 grams total/day) PO dosing: 500 mg BID or 1000 mg daily (depending on the prescribed formulation)
  Vitamin C will be administered through day 56 from start of vitamin C treatment. Patients initially receiving IV administration may be transitioned to PO formulation once tolerating PO intake; per treating physician discretion.

SUMMARY:
After a transplant from another donor, one risk is graft versus host disease (GVHD) that happens because of differences between the donated cells (graft) and the patient's body cells (host). The new cells from the donor might see the body's cells as different and attack them. GVHD can be very serious and cause death. The standard first treatment for GVHD is corticosteroids but not all patients respond and in cases where they don't, they need to go onto other treatments that may or may not be effective. In addition, when GHVD involves the gut it can damage the cells of the gastrointestinal track causing long term problems such as abdominal pain and bowel disturbance. In laboratory studies giving a vitamin C has been able to protect the gastrointestinal cells and help them recover. In this trial the investigators would like to see if vitamin C can do the same thing when given with steroids in patients with GVHD.

The standard first treatment for acute GVHD is corticosteroids but not all patients respond and in cases where they don't, they need to go onto other treatments that may or may not be effective. In addition, when GHVD involves the gut it can damage the cells of the gastrointestinal track causing long term problems such as abdominal pain and bowel disturbance. In the laboratory vitamin C has been able to protect gut stem cells and help them recover and the investigators would like to learn if this happens in people too.

Vitamin C is a readily available supplement. Vitamin C has NOT been approved by the FDA for the treatment of acute GVHD.

DETAILED DESCRIPTION:
Patients enrolled on this trial will receive vitamin C through the vein or by mouth daily for 56 days. This will start at the same time or within 3 days of starting standard treatment for gut GVHD with steroids.

Medical tests before treatment--

Before being treated, patients will receive a series of standard medical tests:

* History and Physical exam
* Blood tests to measure blood cells, kidney and liver function
* A biopsy of the gut to look for GVHD if possible
* Serum pregnancy test for female patients who are of childbearing potential
* An optional stool research sample

Medical tests during and after treatment:

Patients will receive standard medical tests while getting the GVHD treatment and afterwards:

* History and Physical exams
* Monitoring for GVHD
* Blood tests to measure blood cells, kidney and liver function
* A follow-up biopsy of the gut to look for GVHD if possible

To learn more about the way that vitamin C may work on gut stem cells an extra amount of blood will be obtained on the day vitamin C starts, 2 and 4 weeks after starting the vitamin C. The amount of blood taken will be based on the patients weight with up to a maximum of 60 mL (12 teaspoons) of blood to be obtained at any one time. This volume is considered safe but may be decreased if the patient is anemic (have a low red blood cell count).

If patient has a repeat gut biopsy to check GVHD the investigators will request a sample to be used for research purposes.

Patient will receive supportive care for any acute or chronic toxicities, including blood components or antibiotics, and other intervention as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 5 years of age or older at time of enrollment.
2. Patients experiencing their initial presentation of stage 2 or greater acute LGI GVHD (with or without other organ involvement) or stage 1 LGI + skin aGVHD requiring systemic therapy after allogeneic transplant for any malignant or non-malignant indication using any graft/donor source or conditioning intensity.
3. KPS ≥70%
4. Patients should not have received systemic immune suppressive therapy for treatment of active GVHD except for a maximum of 72 hours of steroid therapy (with or without ruxolitinib) prior to enrollment. Topical skin and GI corticosteroids (such as budesonide and oral beclomethasone diproprionate) are allowed.
5. Informed Consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Exclusion Criteria:

1. Relapsed, progressing or persistent malignancy or evidence of minimal residual disease (MRD) requiring withdrawal of systemic immune suppression.
2. Patients with acute GVHD developing after administration of a donor lymphocyte infusion (DLI) for relapse/progression of disease.
3. Patients with uncontrolled infections will be excluded. Infections are considered controlled if appropriate therapy has been instituted and, at the time of enrollment, no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms
4. Known or suspected hypersensitivity to vitamin C.
5. De novo chronic GVHD or overlap syndrome developing before or present at the time of enrollment.
6. Patients receiving other drugs for the treatment of GVHD except as noted above. GVHD prophylaxis agents (e.g., calcineurin inhibitors) may be continued at local Investigator's discretion.
7. Patients on renal replacement therapy.
8. Patients requiring continuous supplemental oxygen > 2L/min to maintain peripheral O2 saturation [SpO2] > 90%.
9. Patients with active hepatic sinusoidal obstructive syndrome (SOS) and/or clinical evidence of impaired hepatic function (ascites or encephalopathy related to liver disease.
10. Patients receiving systemic corticosteroids (CS) for any indication within 7 days before enrollment, except the following:

    1. Corticosteroids administered as premedication for supportive care (such as before transfusion of blood products or before intravenous medications to prevent infusion reactions, fever, etc.).
    2. If steroid therapy has been administered for treatment of a non-GVHD related condition and tapered to < 0.6 mg/kg/day prednisone (0.5 mg/kg/day methylprednisolone) for 7 or more days prior to enrollment.
11. History of G6PD deficiency, sickle cell disease or hemochromatosis.
12. History of oxalate kidney stones.
13. Patients unlikely to be adherent to study specific assessments at the transplant center.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 28 days post-treatment
  The primary endpoint is overall (complete or partial) response to combination of vitamin C with steroids at day 28 post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: LaQuisa Hill, MD, Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: No